CLINICAL TRIAL: NCT06161155
Title: The PROFUN Study: Protein Fermentation Unraveled - Exploring the Relationship Between Digestibility and Metabolite Production.
Brief Title: Protein Fermentation Unraveled (PROFUN) - Exploring the Relationship Between Digestibility and Metabolite Production
Acronym: PROFUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Stichting IMEC-NL (Other)
Responsible Party: Principal Investigator, Guido Hooiveld, Assistant Professor, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL84483.091.23
Record Dates: First submitted 2023-10-19; First posted 2023-12-07 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Protein Fermentation
Keywords: metabolites; dietary protein; digestibility; ingestible

STUDY DESIGN:
Intervention Model Description: After baseline measurements for all participants without dietery intervention, participants will follow a dietary intervention for 7 days followed by a 7-day wash-out period and another 7-day dietary intervention.
Who Masked: Participant
Masking Description: Participants are masked regarding the protein source in the dietary intervention. Participants are not masked regarding the ingestible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein then bovine plasma protein (Active Comparator): During the first dietary intervention, the diet is supplemented with whey protein isolate. During the second dietary intervention, the diet is supplemented with bovine plasma protein.
  Interventions: Combination Product: Protein digestibility
- Bovine plasma protein then whey protein (Active Comparator): During the first dietary intervention, the diet is supplemented with bovine plasma protein. During the second dietary intervention, the diet is supplemented with whey protein isolate.
  Interventions: Combination Product: Protein digestibility

INTERVENTIONS:
Combination Product: Protein digestibility — Two protein sources differing in digestiblity will be used in the dietary intervention to create a difference in protein flow into the large intestine, resulting in different levels of protein fermentation.
  Participants will swallow an ingestible that senses biomarkers related to protein fermentation.

SUMMARY:
Background of the study:

Protein intake is often higher than recommended in Western countries. This leads to increased amounts of protein flowing into the large intestine. Next to increased dietary protein intake, protein digestibility, and endogenous protein losses also affect the amount of protein entering the large intestine. However, these aspects have barely been studied, especially in humans. The large intestine is home to the largest bacterial ecosystem of the body. During the fermentation of protein by these bacteria (microbiota), metabolites are produced such as ammonia, branched-chain fatty acids, biogenic amines, phenolic compounds, indoles, and N-nitroso compounds. There is evidence that some of these metabolites could be harmful for gut epithelia, gastrointestinal health, and health in general after they enter blood circulation. In general, doing measurements inside the gastrointestinal tract is invasive. During this project the protein fermentation will be studied in the gastrointestinal tract using feces and urine, but also in situ using the GISMO GEN1 ingestible. This ingestible contains sensors to measure pH, ammonium, temperature, and redox potential.

Objective of the study:

The primary objectives of this study are:

1. To investigate the feasibility of the GISMO GEN1 System to monitor biomarkers in the gastrointestinal tract by studying the ingestible transit time, data coverage, participant experience, and serious adverse events (if applicable).
2. To study the effect of a 7-day high versus low digestible protein source present in the diet on protein fermentation in healthy subjects, measured by ammonia concentrations.

Study design:

The study is divided into 2 phases. In phase 1, preliminary feasibility of the GISMO GEN1 ingestible system will be assessed and the baseline measurements will be taken without any dietary restrictions. An interim analysis will be performed after phase 1 and only after a positive evaluation of the GISMO GEN1 System, the study will continue with phase 2.

Phase 2 is a randomized cross-over controlled feeding trial. Two diets will be used: one diet containing a high digestible protein source, and the other diet containing a low digestible protein source. Each diet will be given for 7 days, with a wash-out period in between. Measurements done during the dietary interventions will be compared to the other diet, and to the baseline measurements.

Study population:

15 healthy male or female volunteers, age 16 or older, BMI 18.5-30.

Intervention:

A high digestible protein diet (30 g/d whey protein) and a low digestible protein diet (30 g/d bovine plasma protein).

Primary study parameters/outcome of the study:

Ammonia as biomarker for protein fermentation, measured in feces and urine and in situ by the GISMO GEN1 ingestible.

Also, ingestible transit time, data coverage, participant experience, and serious adverse events.

Secundary study parameters/outcome of the study (if applicable):

Secondary study parameters include other protein fermentation related metabolites measured in feces, urine and blood; microbiome composition; transit time; absorption kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age between 16 years or older
* BMI between 18.5-30 kg/m2
* Normal bowel movement: at least one defecation per 48 hours
* Suitable veins for insertion of cannula

Exclusion Criteria:

* Having a current or past medical history or surgical events that may either put the subject as risk because of participation in the study, or influence the results of the study, including, a swallowing disorder, gastrointestinal or liver or endocrine or renal or cardiovascular disease, any other chronic disease, partial bowel resection, renal failure, cancer, nose/throat diseases, gastric bypass surgery, use of anticoagulants; as determined by the medical supervisor;
* Use of any medications in the week before the study that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics, laxatives), or acidity (PPI, H2RA), as determined by medical supervisor;
* Having a bleeding/coagulation disorder, including hemophilia, Von Willebrand disease, Bernard-Soulier, Glanzmann thrombasthenia or thrombocytopenia;
* Swallowing disorders; Among others: dysphagia, any oropharyngeal or oesophageal stricture, functional abnormality, or anxiety disorders related to swallowing disorders;
* Severe dysphagia to food or pills;
* Suspected or known strictures, fistulas, or physiological/mechanical GI obstruction;
* Previous GI abdominal surgery; Except: uncomplicated appendectomy, and/or laparoscopic cholecystectomy;
* Pregnancy, recent childbirth in last 6 months, or actively trying to get pregnant;
* Planned MRI procedure during the study;
* Pacemakers, defibrillator, infusion pump, or other implanted electromedical devices;
* Suffering >2 times per week from: nausea / vomiting / decreased appetite / abdominal pain / high blood pressure / headaches, shakiness, and weakness / fever / diarrhea / constipation;
* Unwilling to undergo an X-ray examination and/or ultrasound (in case sensorcapsule exit cannot be confirmed);
* Working in a professional healthcare facility (e.g. hospital, dental office, emergency room), military area (e.g. submarine, near radar installation), or heavy industrial area (e.g. power plants, automotive, mining, refineries) during the duration of the study;
* Having an allergy or intolerance towards compounds in the prescribed foods (e.g. gluten, lactose, fish, peanuts, soy, nuts);
* Following a vegetarian or vegan diet;
* Use of prebiotic supplements or probiotics for 3 months before the start of the study;
* Use of antibiotics within 2 months of starting the study or planned during the study;
* Excessive alcohol consumption (alcohol: <21 consumptions/week for men, and <14 consumptions/week for women);
* Use of soft drugs within 1 month of starting the study or during the study;
* Use of hard drugs;
* Hemoglobin levels <8.5 mmol/L for men and <7.5 mmol/L for women;
* Participation in another biomedical study;
* Not having a GP;
* Being an employee of Wageningen University, Division of Human Nutrition and Health.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
GISMO GEN1 System feasibility | 3 times approximately 3 days during the trial, within a time frame of 2.5 months
  Ingestible transit time, data coverage, participant experience, and serious adverse events (if applicable)
Ammonia | 3 times during the trial (baseline measurements, dietary intervention 1, dietary intervention 2), within a time frame of 2.5 months
  Ammonia will be measured in feces, urine, and throughout the gastrointestinal tract using the GISMO GEN1 System.

SECONDARY OUTCOMES:
Fermentation related metabolites | 3 times during the trial (baseline measurements, dietary intervention 1, dietary intervention 2), within a time frame of 2.5 months
  Feces, urine, and the GISMO GEN1 ingestible will be used to analyze a range of protein fermentation related metabolites.
pH | 3 times during the trial (baseline measurements, dietary intervention 1, dietary intervention 2), within a time frame of 2.5 months
  pH in feces and measured using the GISMO GEN1 ingestible.
Microbiome composition | 3 times during the trial (baseline measurements, dietary intervention 1, dietary intervention 2), within a time frame of 2.5 months
  Microbiome composition in feces
Transit time | 5 times during the trial (1 times during baseline measurements, twice during dietary intervention 1, twice during dietary intervention 2), within a time frame of 2.5 months
  Transit time measured using the blue dye method, the insoluble marker acid-insoluble-ash, breath analysis, and the GISMO GEN1 ingestible.
Absorption kinetics | 2 times during the trial (dietary intervention 1, dietary intervention 2), within a time frame of 3 weeks
  Amino acid absorption and gut hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided